CLINICAL TRIAL: NCT04694209
Title: Assessment Of Patient Satisfaction and Oral-health Related Quality of Life In Completely Edentulous Patients Receiving Removable Implant Overdentures Versus Fixed Implant Overdentures: A Randomized Clinical Trial
Brief Title: Patient Satisfaction and OHRQoL In Removable Versus Fixed Implant Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iman Abd-ElWahab Radi, PhD (Other)
Responsible Party: Sponsor-Investigator, Iman Abd-ElWahab Radi, PhD, professor of prosthodontics, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151017
Record Dates: First submitted 2020-12-24; First posted 2021-01-05 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Completely Edentulous Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed implant supported prosthesis (Experimental): the prosthesis is an all-on-four prosthesis composed of a hybrid prosthesis. a metal framework, acrylic resin denture base and acrylic resin teeth
  Interventions: Procedure: maxillary and mandibular screw retained hybrid prostheses supported by 4 implants
- Removable implant supported prosthesis (Active Comparator): the prosthesis is an all-on-four prosthesis composed of a telescopic retained overdenture, both primary and secondary copings are custom made. the secondary copings are conncetd via a metal framework
  Interventions: Procedure: maxillary and mandibular telescopic retained overdentures supported by 4 implants

INTERVENTIONS:
Procedure: maxillary and mandibular telescopic retained overdentures supported by 4 implants — The wax of the trial denture was converted into heat-cured acrylic resin using conventional packing and flasking techniques. The prosthesis was finished, polished and screwed in the patient's mouth. Engaging (Internal hex) cylindrical, plastic patterns (Octa plastic cylinder, multi unit abutment, Red, Dentis, Daegu -Korea) were used to construct the primary copings of the telescopic prosthesis.The finished primary copings were scanned using a lab scanner (Shera Echo-scan 7. Dental Wings, Montreal-Canada). This was necessary to design and to mill the wax pattern of the secondary copings using CAD/CAM technology (Dental Wings Software, Dental Wings, Montreal -Canada). Secondary coping was designed to properly fit to the primary coping. The framework was then tried in. At that time it was ready for its intra-oral luting to the secondary copings.
  Arms: Removable implant supported prosthesis
Procedure: maxillary and mandibular screw retained hybrid prostheses supported by 4 implants — Framework of the hybrid prosthesis is waxed using plastic copings attached to multiunit abutments. once the framework is finished , bite is recorded, teeth are set up and the waxed up prosthesis are tried in. IF accepted the wax is eliminated the wax up denture is converted inti heat cured acrylic resin
  Arms: Fixed implant supported prosthesis

SUMMARY:
Objectives to evaluate the oral health-related quality of life and patient satisfaction in completely edentulous patients, when restored by maxillary and mandibular fixed (screw-retained) or removable telescopic retained implant supported prosthesis. 19 patients were randomized to receive either a fixed or a removable maxillary and mandibular full arch implant prosthesis. They were then asked to answer the OHIP-14 and a patient satisfaction questionnaire at 2 weeks, 3, 6 and 12 months post-prosthetic insertion.

DETAILED DESCRIPTION:
Interventions

General operative procedures:

Once the eligibility criteria were fulfilled in a patient, new complete maxillary and mandibular dentures were fabricated for this patient to allow for prosthetically driven implant placement. 4 implants were placed interforaminally so that they were parallel to each other. If the patient had an existing satisfactory denture, that was delivered at least six months ago, it was evaluated for retention, fit, support, stability, occlusion and esthetics. New and old dentures were later used for constructing the scan appliances.

The patients were randomly assigned into two groups with an allocation ratio 1:1. Simple randomization was done by preparing sequentially-numbered, opaque, sealed envelopes, that contained two-times folded cards with the treatment group written inside. Accordingly, the patients were assigned either to group T (control treatment/ telescopic retained implant supported removable overdentures) or group S (test treatment/ screw retained implant supported fixed prosthesis).

The intervention arm : Engaging (Internal hex) cylindrical, plastic patterns (Octa plastic cylinder, multi unit abutment, Red, Dentis, Daegu -Korea) were used to construct the primary copings of the telescopic prosthesis.The finished primary copings were scanned using a lab scanner (Shera Echo-scan 7. Dental Wings, Montreal-Canada). This was necessary to design and to mill the wax pattern of the secondary copings using CAD/CAM technology (Dental Wings Software, Dental Wings, Montreal -Canada). Secondary coping was designed to properly fit to the primary coping. The framework was then tried in. At that time it was ready for its intra-oral luting to the secondary copings.

the control treatment: Once adequate fit of the framework of the hybrid prosthesis was achieved, the wax of the trial denture was converted into heat-cured acrylic resin using conventional packing and flasking techniques. The prosthesis was finished, polished and screwed in the patient's mouth.

Lack of blinding of the operator, the participants and the assessor (patient) due to the obvious dissimilarity between the treatment arms, could have created performance and assessment bias. In an attempt to decrease the performance bias, randomization was delayed until the abutments were connected. When the prosthesis was delivered to the patient, they were requested to answer OHIP-14 and patient satisfaction questionnaires 2 weeks after prosthetic insertion, then 3, 6 and 12 months later.

The aim of this RCT was to evaluate patient satisfaction and oral-health related quality of life in completely edentulous patients receiving removable implant overdentures versus fixed implant hybrid restorations.

Data were statistically described in terms of mean +/- standard deviation (+/- SD), median and range. Comparison of ordinal variables between the study groups was done using Mann Whitney U test for independent samples. Within group comparison of the ordinal data was done using Friedmann test to detect significant differences between time in periods. This was followed by Wilcoxon signed rank test for paired comparisons. Two sided p values less than 0.05 was considered statistically significant. Additionally, a correlation between relevant domains of the OHIP-14 and the patient satisfaction questionnaires was done using Spearman rank correlation test. All statistical calculations were done using computer program IBM SPSS (Statistical Package for the Social Science; IBM Corp, Armonk, NY, USA) release 22 for Microsoft Windows

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous male patients with an age range from 40- 70 years.
2. Patients with a HbA1c equal to or less than 7
3. All patients should have normal maxillo-mandibular relationship (Angle class I).
4. Patients should have maxillary and mandibular ridges at least 7mm in width and 13 mm in height in the interforaminal areas and in the esthetic zones (premolar to premolar regions), respectively. This accommodated a pre-planned implant size of 3.7mm x 10 or 11mm.
5. The maxillary and mandibular ridges should be covered by keratinized attached mucosa at least 5mm in width.
6. An interarch space between the edentulous maxillary and mandibular ridges should not be less than 22 mm to accommodate the planned maxillary and mandibular implant-supported prostheses. This was confirmed by mounted diagnostic casts.
7. Patients who were cooperative and who were psychologically and mentally stable as revealed from the initial interview with the patients were considered eligible.

Exclusion Criteria:

* Females were excluded on purpose to prevent failures associated with osteoporosis and to avoid gender variability which definitely affects the results of patient satisfaction and OHIP.

  2. Patients requiring hard or, soft tissue grafting of the proposed implant sites.

  3. Heavy smokers (more than 10 cigarettes / day) or patients with para-functional habits like clenching or bruxism were excluded. This was important to decrease the risk of implant failure.

  4. Patients with temporo-mandibular joint disorders were considered ineligible because of the expected occlusal disturbances.

  5. Patients with systemic disease that might contra-indicate implants placement or affect osseointegration e.g. uncontrolled diabetes.

  6. Patients who took chemo-or radiotherapy or any drug that might counter-affect the healing process or the quality of bone.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 2 weeks after prosthetic insertion- 1 year
  questionnaire. The patient satisfaction questionnaire is composed of 14 questions concerned with esthetics, speech, mastication, operative and prosthetic procedures, incidence of complications, pre-operative instructions, total time interval, cost, operator, hygienic procedures, overall experience as well as the willingness to repeat or refer others for the procedure.

SECONDARY OUTCOMES:
oral health related quality of life | 2 weeks after prosthetic insertion- 1 year
  OHIP-14 scoring

CONTACTS AND LOCATIONS:
Overall Officials: Amira kheidr, masters, Principal Investigator — Cairo University; Amr El Khadem, phd, Study Director — Cairo University; Samira Ibrahim, phd, Study Chair — Cairo University; Iman Radi, phd, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No